CLINICAL TRIAL: NCT03966105
Title: Prevalence of Amyloidosis in Patients With Lumbar Spinal Stenosis
Brief Title: Prevalence of Wild Type ATTR
Status: Completed | Type: Observational
Sponsor: Oncology Institute of Southern Switzerland (Other)
Collaborators: University of Kiel (Other); Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Adalgisa Condoluci, MD, Resident Physician, Oncology Institute of Southern Switzerland
Other Study IDs: IOSI-EMA-007
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Wild-type Transthyretin Amyloidosis
Keywords: wild-type TTR amyloidosis; lumbar spinal stenosis; prevalence
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with LSS surgery indication
  Interventions: Diagnostic Test: HE and Congo red staining

INTERVENTIONS:
Diagnostic Test: HE and Congo red staining — Biopsies will be formalin fixed, processed routinely, and sent to the Department of Pathology for evaluation by hematoxylin and eosin and Congo red staining by pathologists. Biopsy specimens with confirmed amyloid deposits via Congo red staining will be further analyzed using immunohistochemistry for subtyping.

SUMMARY:
Prospective, observational, single-centre, non-interventional study aiming at reporting the prevalence of ATTRwt in patients with lumbar spinal stenosis (LSS).

DETAILED DESCRIPTION:
The study will include patients that receive surgical management and treatment for LSS, and will consist in the prospective, longitudinal collection of peripheral blood, urine samples, tissue biopsies and clinical data. The results of the project could provide a future benefit for patients with the same condition by: i) identifying accessible and sensitive biomarkers for the identification of patients at risk for having an underlying ATTRwt; ii) optimizing the therapeutic strategies in an era of innovative but cost-intensive treatments; iii) provide the proof of principle for a regular follow-up of patients who eventually will become symptomatic for overt organ ATTRwt involvement; and iv) providing the rationale for future studies based on early access disease-modifying approaches.

ELIGIBILITY:
Inclusion Criteria:

* Male and female ≥ 50 years-old with indication of surgery treatment according to local standards for Lumbar spinal stenosis (LSS) confirmed by MRI
* Availability of the baseline and follow-up annotations
* Informed consent will be obtained from the patient before any study related procedures

Exclusion Criteria:

* Previous diagnosis of amyloidosis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective population of 100 patients undergoing LSS surgery.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Report the prevalence of ATTRwt in patients with CTS and/or LSS. | 2 years
  Prevalence of ATTRwt in a prospective population.

CONTACTS AND LOCATIONS:
Overall Officials: Adalgisa Condoluci, MD, Principal Investigator — Oncology Institute of Southern Switzerland
Locations (1):
- Oncology Institute of Southern Switzerland, Bellinzona, Canton Ticino, Switzerland